CLINICAL TRIAL: NCT06088446
Title: Effect of Intrapulpal Injections on the Post-endodontic Pain in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Intrapulpal Injections on the Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intrapulpal
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementary Intrapulpal injection (Active Comparator): Supplementary Intrapulpal injections were given using a 30-gauze needle with sufficient back pressure.
  Interventions: Procedure: Supplementary anesthetic injections
- Intraligamentary injection (Active Comparator): Intraligamentary injections were given using an intraligamentary syringe with back-pressure after a failed primary inferior alveolar nerve block.
  Interventions: Procedure: Supplementary anesthetic injections

INTERVENTIONS:
Procedure: Supplementary anesthetic injections — Supplementary anesthetic injections after failed primary nerve block

SUMMARY:
To achieve painless treatment in patients with a failed primary IANB, supplementary anesthesia has been advised. The majority of the studies evaluating intrapulpal injections have been performed on asymptomatic teeth. Very limited research has been dedicated to the evaluation of different variables in intrapulpal injections in patients with symptomatic irreversible pulpitis. The aim of this study was to evaluate postoperative pain after an intrapulpal anesthesia injection given after a failed inferior alveolar nerve block (IANB), in patients with symptomatic irreversible pulpitis. This prospective, randomized, double-blind clinical trial was carried out at the Department of Conservative Dentistry and Endodontics, Faculty of Dentistry, Jamia Millia Islamia. One hundred and eight adult patients, with symptomatic irreversible pulpits in a mandibular first or second molar received an initial IANB with 2% lidocaine. Pain during the endodontic treatment was assessed using a visual analog scale (VAS). Patients experiencing pain on endodontic intervention were randomly allocated to one of the two treatment groups: one group received a supplementary intrapulpal injection while the other received a supplementary intraligamentary injection The presence of postoperative pain was assessed at 1, 2, 3, and 7 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic carious exposed mandibular first or second molars.
* Positive and prolonged response to thermal sensitivity tests and electric pulp tests.
* Vital coronal pulp on access cavity preparation.
* American Society of Anesthesiologists class I or II medical history.
* Ability to understand the use of pain scales.

Exclusion Criteria:

* Active pain in more than 1 tooth.
* Teeth with fused roots.
* Radiographic evidence of an extra root.
* Large restorations with overhanging margins.
* Full crowns or deep periodontal pockets.
* Known allergy or contraindications to any content of the local anesthetic solution or NSAIDs
* History of known or suspected drug abuse.
* Taking any drugs which could affect the pain perception, e.g, opiods, antidepressants, anticonvulsants, muscle relaxants, anxiolytics, sedatives, nsaids. 23
* Pregnant or breastfeeding patients.
* Patients with asthma, gastric ulcers, and bleeding disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Post-endodontic pain using a visual analouge scale (VAS) | 6hours, 1 day, 3 days, 7 days
  Evaluation of numerical visual analouge pain scores after the completion of root canal treatment. The scale was 170mm long and the the values were continous and numerical. The 0 indicates no pain and 170 indicates the maximum possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Jamia MIliia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided